CLINICAL TRIAL: NCT05818579
Title: The Effects of Therapeutic Virtual Reality Experience to Promote Mental Well-being in Older People Living With Physical Disabilities in Long-term Care Facilities
Brief Title: Virtual Reality for Mental Well-being in Older People With Physical Disabilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tung Wah College (Other)
Collaborators: Chinese University of Hong Kong (Other); Golden Age Foundation (Unknown); Pok Oi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHI2_0071
Record Dates: First submitted 2023-04-05; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Mental Health Wellness 1; Physical Disability
Keywords: Mental wellbeing; Virtual reality; Physical disability; Older people

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In the proposed study, only the outcome assessor will be blinded to the group labels. Participants and interventionists are impossible to be blinded in this study. The group labels will not be known to the outcome assessors and will not appear on any documents that the outcome assessors can access. The participants, family members, and staff members of the LTCF are prohibited to disclose the group labels of the participants to the outcome assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): The investigators will administer a virtual reality experience programme to promote mental wellbeing of the participants
  Interventions: Other: Virtual reality experience
- Usual care (No Intervention): The investigators will not provide any interventions to the participants.

INTERVENTIONS:
Other: Virtual reality experience — The VR experience is launched on the participants using all-in-one VR head-mount devices. Tablet computers are used to optimize the settings by the intervention facilitators. Each session lasts for approximately one hour with 10 minutes spent on the briefing, 20 minutes spent on the VR experience, and 30 minutes spent on the post-VR group discussion. There are two sessions per week. The whole course lasts for six weeks and there are a total of 12 sessions.
  Arms: Virtual reality

SUMMARY:
Objectives This study aims to examine the effects of the therapeutic virtual reality (VR) experience in older people with physical disabilities in long-term care facilities (LTCF) in 1) increasing mental well-being, 2) reducing depressive symptoms, 3) reducing loneliness, 4) increasing health-related quality of life, and 5) increasing perceived social support. If this intervention is successful, this study will yield new knowledge about the effects of this innovative intervention. Also, an innovative VR intervention will be available to promote the mental well-being of older residents in LTCF.

Trial design This study employs a single-blinded, two-parallel-group (intervention-to-control group ratio=1:1), non-inferiority, randomized controlled trial.

Study setting This study will be conducted in the LTCF. Participants will be recruited from Care & Attention Homes for the Elderly and Nursing Homes under the governance of the Social Welfare Department in Hong Kong.

Eligibility criteria Inclusion: 1) Aged 60 years or above; 2) LTCF residents; and 3) Physical disability, defined as the Modified Barthel Index (MBI) score of ≤ 90 (i.e., moderately dependent or worse). Exclusion: 1) Probably dementia, as defined by a Montreal Cognitive Assessment score of < 20, 2) Severe visual impairment, as defined by a lens-corrected visual acuity score of < 6/60, 3) Severe hearing impairment, as defined by failed whispered voice test, 4) Bilateral upper limb paralysis, as defined by the Medical Research Council Muscle Power Scale of < 4, or 5) Participated in any VR activities in the past six months or concurrently.

Consent All participants will be asked to give their written informed consent to participate in the proposed study.

Groups Participants allocated to the intervention group will participate in the 6-week VR experience programme. Participants allocated to the control will receive the usual care provided by the LTCF, such as personal care, regular basic medical and nursing care, and social support, as committed by the Social Welfare Department. The participants allocated to the intervention group receive the same usual care provided by the LTCF. The research team does not interfere with the services provided to the participants in either group.

Outcomes Demographic data including age, gender, level of education, number of chronic illnesses, length of stay in the LTCF, and experience of participation in VR activities will be collected. Outcomes include mental well-being, depressive symptoms, loneliness, health-related quality of life, and perceived social support.

Participant timeline Potential participants will be recruited in the phase of Enrolment, in which the eligibility screen and informed consent will be implemented. Then, in the phase of the Pre-treatment Assessment (i.e., T0,), demographic and outcome data will be collected. Subsequently, in the phase allocation, participants will be randomly allocated to either the therapeutic virtual reality experience group or the control group. Then, interventions will be implemented. In the phase of the Post-treatment Assessment (i.e., T1), outcome data will be collected once again.

Analysis methods Demographic and outcome data collected at baseline will be reported either as means with standard deviation or as frequencies with percentages according to their levels of measurement as a whole sample and by groups. Generalized estimating equations (GEE) will be employed to separately test the hypothesis on the five outcomes as dependent variables (i.e., mental well-being, depressive symptoms, loneliness, health-related quality of life, perceived social support), The independent variables will be the same across all GEEs: group (two categories: intervention and control groups), timepoint (two categories: T0 and T1), and group x timepoint. The primary interpretation of the results will be based on the intention-to-treat analysis without adjusting for covariates. The level of significance will be set at 0.05. Missing data will be managed following a practical guide with flowcharts using various methods (e.g., multiple imputation, single imputation, or no imputation).

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or above;
* LTCF residents; and
* Physical disability, defined as the Modified Barthel Index (MBI) score of ≤ 90 (i.e., moderately dependent or worse).

Exclusion Criteria:

* Probably dementia, as defined by a Montreal Cognitive Assessment (MoCA) score of < 20,
* Severe visual impairment, as defined by a lens-corrected visual acuity score of < 6/60,
* Severe hearing impairment, as defined by failed whispered voice test.
* Bilateral upper limb paralysis, as defined by the Medical Research Council Muscle Power Scale of < 4. or
* Participated in any virtual reality activities in the past six months or concurrently.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2025-02-14 (Estimated); Study Completion 2025-05-14 (Estimated)

PRIMARY OUTCOMES:
Mental well-being | 6 weeks
  The World Health Organization Five Well-being Index will be used to measure mental well-being.

SECONDARY OUTCOMES:
Depressive symptoms | 6 weeks
  The 9-item Patient Health Questionnaire will be used to measure depressive symptoms over the past two weeks.
Loneliness | 6 weeks
  The Chinese version of the 6-item De Jong Gierveld Loneliness Scale will be used to measure loneliness.
Health-related quality of life | 6 weeks
  The Hong Kong version of the EuroQol 5-dimensions instrument with a five-level scale will be used to measure health-related quality of life.
Perceived social support | 6 weeks
  The Chinese version of the Multiple Scale of Perceived Social Support (MSPSS) will be used to measure perceived social support.

IPD SHARING:
Plan to Share IPD: Undecided
The data will be provided upon request.

REFERENCES:
- [Derived] Kwan RYC, Ng F, Lam LCW, Yung RC, Sin OSK, Chan S. The effects of therapeutic virtual reality experience to promote mental well-being in older people living with physical disabilities in long-term care facilities. Trials. 2023 Aug 26;24(1):558. doi: 10.1186/s13063-023-07592-7. PMID 37633916